CLINICAL TRIAL: NCT04266301
Title: A Randomized, Double-blind, Placebo-controlled Phase III Multi-center Study of Azacitidine With or Without MBG453 for the Treatment of Patients With Intermediate, High or Very High Risk Myelodysplastic Syndrome (MDS) as Per IPSS-R, or Chronic Myelomonocytic Leukemia-2 (CMML-2)
Brief Title: Study of Efficacy and Safety of MBG453 in Combination With Azacitidine in Subjects With Intermediate, High or Very High Risk Myelodysplastic Syndrome (MDS) as Per IPSS-R, or Chronic Myelomonocytic Leukemia-2 (CMML-2)
Acronym: STIMULUS-MDS2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: In December 2023, Novartis decided to terminate the sabatolimab clinical development program early after Phase II (MDS1) and Phase III (MDS2) studies failed to meet their primary objectives. The termination was not due to safety concerns.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMBG453B12301; 2019-002089-11 (EudraCT Number)
Record Dates: First submitted 2020-01-21; First posted 2020-02-12 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic
Keywords: MBG453; Phase III; TIM-3; azacitidine; myelodysplastic syndrome; MDS; chronic myelomonocytic leukemia; CMML-2; Sabatolimab; high or; very high risk myelodysplastic syndrome; Chronic Myelomonocytic Leukemia-2
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — sabatolimab; Azacitidine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sabatolimab (MBG453) + Azacitidine (Experimental): Participants received sabatolimab plus Azacitidine
  Interventions: Drug: Sabatolimab; Drug: Azacitidine
- Placebo + Azacitidine (Placebo Comparator): Participants received placebo plus Azacitidine.
  Interventions: Drug: Azacitidine; Drug: Placebo

INTERVENTIONS:
Drug: Sabatolimab — A dose of MBG453 800 mg was administered intravenously (IV) every 4 weeks (Q4W).
  Other Names: MBG453
  Arms: Sabatolimab (MBG453) + Azacitidine
Drug: Azacitidine — A dose of Azacitidine 75 mg/m2 was administered IV or subcutaneously (SC) on Day 1-7, or Day 1-5, 8 and 9.
Drug: Placebo — A dose of placebo 800 mg was administered intravenously every 4 weeks (Q4W).
  Arms: Placebo + Azacitidine

SUMMARY:
This was a Phase III multi-center, randomized, two-arm parallel-group, double-blind, placebo-controlled study of MBG453 or placebo added to azacitidine in adult participants with intermediate, high or very high-risk myelodysplastic syndrome (MDS) as per IPSS-R, or Chronic Myelomonocytic Leukemia-2 (CMML-2) who are not eligible for intensive chemotherapy or hematopoietic stem cell transplantation (HSCT) according to medical judgment by the investigator.

The purpose of the current study was to assess clinical effects of MBG453 in combination with azacytidine in adult participants with IPSS-R intermediate, high, very high risk MDS and CMML-2.

DETAILED DESCRIPTION:
This was a Phase III multi-center, randomized, two-arm parallel-group, double-blind, placebo-controlled study of MBG453 or placebo added to azacitidine in adult participants with intermediate, high or very high-risk myelodysplastic syndrome (MDS) as per IPSS-R, or Chronic Myelomonocytic Leukemia-2 (CMML-2).

The primary objective of this study was to compare overall survival (OS) in the MBG453 plus azacitidine arm versus placebo plus azacitidine arm where OS was the time from randomization until death due to any cause.

Participants were randomized in a 1:1 ratio to treatment arms as follow: MBG453 800 mg IV Q4W plus azacitidine, Placebo IV Q4W plus azacitidine.

The randomization was stratified into 4 groups: intermediate risk MDS, high risk MDS, very high risk MDS and CMML-2.

All participants who discontinued both study treatments were to have entered a long-term post-treatment follow-up including response and PRO assessments, and/or survival follow-up for up to 5 years after the last participant was randomized.

Participants were receiving treatment until they experienced progression of disease (including transformation to acute leukemia per WHO 2016 classification), experienced unacceptable toxicity or discontinued the study treatment for other reasons.

Continuation of study treatment beyond progression (excluding transformation to acute leukemia: continuation in this case was not possible) could have been possible in selected participants.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study
* Age ≥ 18 years at the date of signing the informed consent form
* Morphologically confirmed diagnosis of myelodysplastic syndrome (MDS) based on WHO 2016 classification (Arber et al 2016) by local investigator assessment with one of the following Prognostic Risk Categories, based on the revised International Prognostic Scoring System (IPSS-R):

  * Very high (> 6 points)
  * High (> 4.5 - ≤ 6 points)
  * Intermediate (> 3 - ≤ 4.5 points) Or Morphologically confirmed diagnosis of Chronic Myelomonocytic Leukemia -2 based on WHO 2016 classification (Arber et al 2016, including persistent monocytosis) by local investigator assessment with WBC < 13 x 109/L at time of initial diagnosis
* Indication for azacitidine treatment according to the investigator, based on local standard medical practice and institutional guidelines for treatment decisions
* Not eligible at time of screening for intensive chemotherapy according to the investigator, based on local standard medical practice and institutional guidelines for treatment decisions, including assessment of individual clinical factors such as age, comorbidities and performance status
* Not eligible at time of screening for hematopoietic stem cell transplantation (HSCT) according to the investigator, based on local standard medical practice and institutional guidelines for treatment decisions, including assessment of individual clinical factors such as age, comorbidities, performance status, and donor availability
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2

Exclusion Criteria:

* Prior exposure to TIM-3 directed therapy at any time. Prior therapy with immune checkpoint inhibitors (e.g, anti-CTLA4, anti-PD-1, anti-PD-L1, or anti-PD-L2), cancer vaccines is allowed except if the drug was administered within 4 months prior to randomization
* Previous first-line treatment for intermediate, high, very high risk myelodysplastic syndromes (based on IPSS-R) or CMML with any antineoplastic agents including for example chemotherapy, lenalidomide and hypomethylating agents (HMAs) such as decitibine and azacitidine. However, previous treatment with hydroxyurea or leukopheresis to reduce WBC count is allowed prior to randomization.
* Investigational treatment received within 4 weeks or 5 half-lives of this investigational treatment, whatever is longer, prior to randomization. In case of a checkpoint inhibitor: a minimal interval of 4 months prior to randomization is necessary to allow randomization.
* Subjects with Myelodysplastic syndrome (MDS) based on 2016 WHO classification (Arber et al 2016) with revised International Prognostic Scoring System (IPSS-R) ≤ 3
* Diagnosis of acute myeloid leukemia (AML) including acute promyelocytic leukemia and extra-medullary acute myeloid leukemia, primary or secondary myelofibrosis based on WHO 2016 classification (Arber et al 2016)
* Diagnosis of therapy related myeloid neoplasms based on WHO 2016 classification (Arber et al 2016)
* History of organ or allogeneic hematopoietic stem cell transplant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (134):
- United States (11):
  - Yuma Regional Cancer Center, Yuma, Arizona
  - University of California LA, Los Angeles, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University Of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hackensack University Medical Ctr, Hackensack, New Jersey
  - Weill Cornell Medicine NY-Presb, New York, New York
  - University of Rochester Medical Ctr, Rochester, New York
  - University of Virginia, Charlottesville, Virginia
- Novartis Investigative Site, Pilar, Buenos Aires, Argentina
- Australia (3):
  - Novartis Investigative Site, Wooloongabba, Queensland
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Perth, Western Australia
- Austria (3):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
- Belgium (2):
  - Novartis Investigative Site, Roeselare, West-Vlaanderen
  - Novartis Investigative Site, Brasschaat
- Brazil (2):
  - Novartis Investigative Site, Florianópolis, Santa Catarina
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (2):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Toronto, Ontario
- Novartis Investigative Site, Viña del Mar, Región de Valparaíso, Chile
- China (11):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shenzhen, Guangdong
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Jinan
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Colombia (2):
  - Novartis Investigative Site, Rionegro, Antioquia
  - Novartis Investigative Site, Bogotá
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Prague
- Finland (2):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Kuopio
- France (6):
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (9):
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Velbert, North Rhine-Westphalia
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Ulm
- Greece (2):
  - Novartis Investigative Site, Alexandroupoli
  - Novartis Investigative Site, Pátrai
- India (5):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Faridabad, Haryana
  - Novartis Investigative Site, Madurai, Tamil Nadu
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Delhi
- Israel (2):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Tel Aviv
- Italy (8):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Roma, RM
- Japan (11):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Yamagata, Yamagata
  - Novartis Investigative Site, Osaka
- Novartis Investigative Site, Beirut, Lebanon
- Novartis Investigative Site, Vilnius, Lithuania
- Malaysia (4):
  - Novartis Investigative Site, George Town, Pulau Pinang
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Kuala Lumpur
  - Novartis Investigative Site, Kuala Selangor
- Mexico (4):
  - Novartis Investigative Site, Satélite, Edo Mexico
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Morelia, Michoacán
  - Novartis Investigative Site, Estado de México
- Novartis Investigative Site, Groningen, Provincie Groningen, Netherlands
- Novartis Investigative Site, Khoudh, Oman
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Novartis Investigative Site, Saint Petersburg, Russia
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Singapore, Singapore
- South Korea (3):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seoul
  - Novartis Investigative Site, Seoul
- Spain (7):
  - Novartis Investigative Site, Badalona, Barcelona
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Switzerland (2):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Zurich
- Taiwan (6):
  - Novartis Investigative Site, Hualien City
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Liouying Township
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Thailand (4):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Samsun, Atakum
  - Novartis Investigative Site, Edirne, Merkez
  - Novartis Investigative Site, Istanbul, Pendik
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Izmir
- United Kingdom (4):
  - Novartis Investigative Site, Portsmouth, Hants
  - Novartis Investigative Site, Edinburgh, Scotland
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of participants who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Zeidan AM, Giagounidis A, Sekeres MA, Xiao Z, Sanz GF, Hoef MV, Ma F, Hertle S, Santini V. STIMULUS-MDS2 design and rationale: a phase III trial with the anti-TIM-3 sabatolimab (MBG453) + azacitidine in higher risk MDS and CMML-2. Future Oncol. 2023 Mar;19(9):631-642. doi: 10.2217/fon-2022-1237. Epub 2023 Apr 21. PMID 37083373
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2874

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study randomized participants in 149 centers in 36 participating countries.
Groups:
- Sabatolimab (MBG453) + Azacitidine: Participants were randomized to sabatolimab plus Azacitidine
- Placebo + Azacitidine: Participants were randomized to placebo plus Azacitidine
Period: Overall Study
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Started | 265 | 265
Participants Treated | 264 | 264
Participants Not treated | 1 | 1
Discontinued from treatment | 264 | 264
Entered post-treatment | 68 | 71
Did not enter post-treatment | 196 | 193
Discontinued from study | 265 | 265
Full Analysis See (FAS) | 265 | 265
Safety Set (Two participants (one per arm) did not receive treatment and were excluded from the Safety Set. One sabatolimab-assigned participant withdrew consent pre-treatment. Another, randomized to placebo, progressed to AML before treatment and died. One sabatolimab-assigned participant progressed to AML, received only azacitidine, and was analyzed in the placebo Safety Set.) | 263 | 265
Completed (Completed = Completed treatment) | 0 | 0
Not Completed | 265 | 265
Not completed — Progressive Disease | 111 | 92
Not completed — Adverse Event | 41 | 43
Not completed — Death | 26 | 35
Not completed — Hematopoietic Stem-Cell Transplantation (HSCT) Planned | 22 | 22
Not completed — Study Terminated by Sponsor | 22 | 27
Not completed — Participant Decision | 22 | 28
Not completed — Physician Decision | 14 | 9
Not completed — New Therapy for Study Indication | 2 | 4
Not completed — Protocol Deviation | 2 | 4
Not completed — Guardian Decision | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Participants Not Treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) comprised of all participants to whom study treatment had been assigned by randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine | Total
Number analyzed (Participants) | 265 | 265 | 530
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.2 (11.46) | 69.1 (11.23) | 69.6 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 79 | 183
  Male | 161 | 186 | 347
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 150 | 134 | 284
  Asian | 111 | 124 | 235
  Black or African American | 3 | 4 | 7
  American Indian or Alaska Native | 1 | 2 | 3
  Unknown | 0 | 1 | 1
ECOG performance status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status scale is a widely used standard of care criteria used to assess the functional status of a patient with cancer to measure how the disease impacts the patient's daily living abilities. This scale has a range from 0 - 5. The higher the grade, the worse the patient's abilities: 0 implies fully active, able to carry on all pre-disease performance without restriction and 5 implies death.
  Participants
    ECOG performance status: 0 | 92 | 101 | 193
    ECOG performance status: 1 | 161 | 141 | 302
    ECOG performance status: 2 | 12 | 23 | 35

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) (Primary Efficacy Results)
Description: OS is the time from randomization until death due to any cause.
Time Frame: up to approx. 39 months
Population: FAS comprised of all participants to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 265 | 265
Months | 22.31 [19.55 to 24.74] | 18.83 [15.38 to 23.72]
Statistical Analysis 1: Comparison: Sabatolimab (MBG453) + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; p = 0.0825, Log Rank — P Value is 1-sided; Log-rank test stratified by randomization stratification factor (Intermediate risk MDS, High risk MDS, Very high risk MDS, CMML-2) as per IRT; Hazard Ratio (HR) = 0.847, 95% CI 2-sided [0.671 to 1.070]

2. Primary Outcome: Overall Survival (OS) (Final Efficacy Results)
Description: OS is the time from randomization until death due to any cause.
Time Frame: up to approx. 52 months
Population: FAS comprised of all participants to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 265 | 265
Months | 22.18 [19.55 to 24.41] | 18.83 [15.38 to 23.72]
Statistical Analysis 1: Comparison: Sabatolimab (MBG453) + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; Hazard Ratio (HR) = 0.863, 95% CI 2-sided [0.693 to 1.076]

3. Secondary Outcome: Key Secondary Endpoint 1: Time to Definitive Deterioration of Fatigue Using Functional Assessment of Cancer Therapy (FACIT)-Fatigue Score
Description: FACIT-Fatigue score is a 13-item questionnaire designed to assess fatigue in cancer participants. All items use a 5-point scale ranging from 0 to 4 (0=Not at All to 4=Very Much). The total score ranges from 0 to 52 with higher values representing better quality of life. Time to definitive deterioration of fatigue is defined as time from randomization to at least 3 points worsening from baseline in FACIT-fatigue scores with no subsequently observed improvement above this threshold, or death due to any cause, whichever occurred first.
Time Frame: up to approx. 52 months
Population: FAS comprised of all participants to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 265 | 265
Months | 13.37 [11.96 to 15.90] | 11.76 [10.15 to 13.86]
Statistical Analysis 1: Comparison: Sabatolimab (MBG453) + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; p = 0.2132, Log Rank — P Value is 1-sided; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.921, 95% CI 2-sided [0.750 to 1.130]

4. Secondary Outcome: Key Secondary Endpoint 2: Red Blood Cell (RBC) Annualized Transfusion Free Rate for Transfusion
Description: Annualized transfusion free rate is defined as the average number of days in RBC transfusion-free intervals in a year (i.e., the total number of days in RBC transfusion-free intervals divided by the total days in the study multiplied by 365.25), where RBC transfusion-free intervals correspond to cumulative times of intervals with no evidence of RBC transfusion for at least 8 weeks at any point after randomization until death due to any cause.
Time Frame: up to approx. 52 months
Population: FAS comprised of all participants to whom study treatment had been assigned by randomization.
Measure: Median (Full Range); unit: days per year
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 265 | 265
days per year | 184.3 [0 to 365] | 175.7 [0 to 365]
Statistical Analysis 1: Comparison: Sabatolimab (MBG453) + Azacitidine; Test type: Superiority; p = 0.4692, negative binomial regression model — P Value is 1-sided; negative binomial regression model with log link stratified by randomization stratification factor as per IRT and baseline transfusion status

5. Secondary Outcome: Key Secondary Endpoint 3: Percentage of Participants With at Least 3 Point Confirmed Improvement From Baseline in FACIT-fatigue Scores
Description: FACIT-Fatigue score is a 13-item questionnaire designed to assess fatigue in cancer participants. All items use a 5-point scale ranging from 0 to 4 (0=Not at All to 4=Very Much). The total score ranges from 0 to 52 with higher values representing better quality of life. The responder is defined as having 3 points improvement from baseline confirmed by a second improvement of 3 points at any time, regardless of preceding worsening. A participant who could not improve was considered as a non-responder.
Time Frame: up to approx. 52 months
Population: FAS comprised of all participants to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants with response
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 265 | 265
Percentage of participants with response | 39.6 [33.7 to 45.8] | 40.8 [34.8 to 46.9]
Statistical Analysis 1: Comparison: Sabatolimab (MBG453) + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; p = 0.4865, Cochran-Mantel-Haenszel — P Value is 1-sided; exact CMH Chi-square statistic, adjusting for randomization stratification factor as per IRT; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.7 to 1.4]

6. Secondary Outcome: Key Secondary Endpoint 4: Percentage of Participants With at Least 10 Point Confirmed Improvement From Baseline in Physical Functioning Using European Organization for Research and Treatment of Cancer's Core Quality of Life Questionnaire (EORTC QLQ-C30)
Description: EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer participants. Participants' responses to 5 questions about their physical functioning (Items 1-5) are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A high score indicates a high / healthy level of functioning. The responder is defined as having 10 points improvement from baseline confirmed by a second improvement of 10 points at any time, regardless of preceding worsening. A participant who could not improve was considered as a non-responder.
Time Frame: up to approx. 52 months
Population: FAS comprised of all participants to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants with response
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 265 | 265
Percentage of participants with response | 30.2 [24.7 to 36.1] | 22.6 [17.7 to 28.2]
Statistical Analysis 1: Comparison: Sabatolimab (MBG453) + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; p = 0.5743, Cochran-Mantel-Haenszel — P Value is 1-sided; exact CMH Chi-square statistic, adjusting for randomization stratification factor as per IRT; Odds Ratio (OR) = 1.48, 95% CI 2-sided [1 to 2.2]

7. Secondary Outcome: Key Secondary Endpoint 5: Percentage of Participants With at Least 10 Point Confirmed Improvement From Baseline in Emotional Functioning Using EORTC-QLQ-C30
Description: EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer participants. Participants' responses to 4 questions about their emotional functioning (Items 21-24) are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A high score indicates a high / healthy level of functioning. The responder is defined as having 10 points improvement from baseline confirmed by a second improvement of 10 points at any time, regardless of preceding worsening. A participant who could not improve was considered as a non-responder.
Time Frame: up to approx. 52 months
Population: FAS comprised of all participants to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 265 | 265
Percentage of participants | 31.7 [26.1 to 37.7] | 28.3 [23.0 to 34.1]
Statistical Analysis 1: Comparison: Sabatolimab (MBG453) + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; p = 0.2126, Cochran-Mantel-Haenszel — P Value is 1-sided; exact CMH Chi-square statistic, adjusting for randomization stratification factor as per IRT; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.8 to 1.7]

8. Secondary Outcome: Percentage of Participants With Either CR, or mCR, or PR, or HI in Each Treatment Arm According to International Working Group for MDS (IWG-MDS) as Per Investigator Assessment
Description: Response rate of participants with complete remission (CR), or marrow remission (mCR), or partial remission (PR), or hematologic improvement (HI).
  CR: where the Bone marrow: ≤ 5% blasts with normal maturation of all cell lineages and Peripheral blood: where Hgb ≥ 10 g/dL AND Platelets ≥ 100*109/L AND Neutrophils ≥ 1.0*109/L AND Peripheral blasts 0%.
  mCR: Bone marrow: ≤ 5% blasts and blast count decrease by ≥ 50% compared to baseline; Peripheralblood/transfusion: Marrow CR may be achieved with or without improved blood counts or with or without transfusions PR: All CR criteria except bone marrow: ≥50% decrease from baseline in blasts in bone marrow AND blast count in bone marrow >5%.
  HI: restoration or enhancement of the function of the body's blood cell-producing system that must last as least 8 weeks.
Time Frame: up to approx. 52 months
Population: FAS comprised of all participants to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 265 | 265
Percentage of participants | 58.1 [51.9 to 64.1] | 47.5 [41.4 to 53.7]

9. Secondary Outcome: Percentage of Participants With Stable Disease (SD) According to International Working Group for MDS (IWG-MDS) as Per Investigator Assessment
Description: Response rate of participants with stable disease. SD is the failure to achieve at least partial response (PR), but no evidence of progression for >8 weeks.
Time Frame: up to approx. 52 months
Population: FAS comprised of all participants to whom study treatment had been assigned by randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 265 | 265
Percentage of participants | 20.0 | 19.6

10. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization to disease progression (including transformation to acute leukemia per WHO 2016), relapse from CR (IWG-MDS), or death. Disease progression: bone marrow blasts increase ≥ 50% over baseline, to > 5% if initially < 5%, > 10% if 5%-<10%, or > 20% if 10%-<20%. Includes a peripheral blood count decrease ≥ 50% from maximum remission/response levels: neutrophils < 1.0x109/L, platelets < 100x109/L, or hemoglobin drop ≥ 2 g/dL to < 10 g/dL, becoming transfusion-dependent.
  Relapse from CR: baseline bone marrow blast % return, neutrophils decrease ≥ 50% to < 1.0x109/L, platelets decrease ≥ 50% to < 100x109/L, or hemoglobin drop ≥ 1.5 g/dL to < 10 g/dL, becoming transfusion-dependent.
  Leukemia transformation: > 20% blasts per WHO 2016 (Arber et al 2016).
Time Frame: up to approx. 52 months
Population: FAS comprised of all participants to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 265 | 265
Months | 14.26 [12.22 to 17.74] | 10.12 [8.64 to 11.14]
Statistical Analysis 1: Comparison: Sabatolimab (MBG453) + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; Hazard Ratio (HR) = 0.710, 95% CI 2-sided [0.576 to 0.875]

11. Secondary Outcome: Leukemia-free Survival (LFS)
Description: LFS is defined as the time from randomization to ≥ 20% blasts in bone marrow/peripheral blood (per WHO 2016 classification) or diagnosis of extramedullary acute leukemia, or death due to any cause
Time Frame: up to approx. 52 months
Population: FAS comprised of all participants to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 265 | 265
Months | 19.84 [17.15 to 24.21] | 13.73 [11.79 to 18.73]
Statistical Analysis 1: Comparison: Sabatolimab (MBG453) + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; Hazard Ratio (HR) = 0.815, 95% CI 2-sided [0.640 to 1.038]

12. Secondary Outcome: Number of Participants Who Become Red Blood Cells (RBC) Transfusion Independent After Randomization
Description: Improvement in RBC transfusion independence as per International Working Group for MDS (IWG-MDS) criteria. RBC transfusion independence was defined as having received 0 units of RBC transfusions during at least 8 consecutive weeks after randomization. The number of participants was shown in only those with transfusion dependence at baseline (BL).
Time Frame: up to approx. 52 months
Population: Participants of the full analysis set (FAS) who were RBC transfusion dependent at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 96 | 108
Participants | 50 | 53

13. Secondary Outcome: Number of Participants Who Become Platelets Transfusion Independent After Randomization
Description: Improvement in Platelets transfusion independence as per International Working Group for MDS (IWG-MDS) criteria. Platelets transfusion independence was defined as having received 0 units of Platelets transfusions during at least 8 consecutive weeks after randomization. The number of participants was shown in only those with transfusion dependence at baseline (BL).
Time Frame: up to approx. 52 months
Population: Participants of the full analysis set (FAS) who were Platelets transfusion dependent at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 23 | 28
Participants | 11 | 10

14. Secondary Outcome: Pharmacokinetics of MBG453 (Parameter Cmax)
Description: Cmax is the maximum (peak) observed drug concentration after single dose administration (mass x volume-1).
Time Frame: 0 hr (pre-dose) & 2 hrs (post-dose) of Cycle (C) 1 Day (D) 8 and 0 hr (pre-dose) & 2 hrs (post-dose) of C3D8
Population: Pharmacokinetic Analysis Set (PAS) included all participants in the Safety Set, who had at least one evaluable PK concentration.
  Safety Set included all participants who received at least one dose of any component of the study treatment, and they were analyzed according to the study treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/ml
Groups:
- Sabatolimab (MBG453): Participants received sabatolimab.
Arm/Group | Sabatolimab (MBG453)
Number analyzed (Participants) | 8
ug/ml
  Cycle 1 | 232 (20.9)
  Cycle 3: number analyzed (Participants) | 6
  Cycle 3 | 239 (39.5)

15. Secondary Outcome: Pharmacokinetics of MBG453 (Parameter AUC)
Description: AUCinf is the AUC from time zero to infinity (mass x time x volume-1).
Time Frame: 0 hr (pre-dose) & 2 hrs (post-dose) of Cycle (C) 1 Day (D) 8 and 0 hr (pre-dose) & 2 hrs (post-dose) of C3D8
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/ml
Arm/Group | Sabatolimab (MBG453)
Number analyzed (Participants) | 4
day*ug/ml
  Cycle 1 | 2670 (45.9)
  Cycle 3: number analyzed (Participants) | 3
  Cycle 3 | 4930 (1.5)

16. Secondary Outcome: ADA Prevalence at Baseline and ADA-positive Participants On-treatment
Description: Anti-drug Antibody (ADA) prevalence is the number of participants with at least one sample meeting the criteria at baseline. ADA-positive participants were calculated as the number of participants with at least one on-treatment ADA-positive sample divided by the number of participants with a determinant baseline IG sample and at least one determinant post-baseline IG sample.
Time Frame: Baseline, up to approx. 39 months
Population: Immunogenicity Incidence Set includes all participants in the Immunogenicity prevalence set with a non-missing baseline ADA sample and at least one non-missing post-baseline ADA sample.
  The Immunogenicity prevalence set includes all participants in the Safety Set with a non-missing baseline ADA sample or at least one non-missing post-baseline ADA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Sabatolimab (MBG453)
Number analyzed (Participants) | 249
Participants
  ADA prevalence (i.e., ADA positive) at baseline | 24
  ADA-positive participants on-treatment | 34

17. Secondary Outcome: Change From Baseline in the European Quality of Life (EuroQol) - 5 Dimensions, 5 Level Questionnaire (EQ-5D-5L) Score Over Time
Description: The EQ-5D-5L comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. For each of the 5 dimensions, subject's responses are scored on a 5-point scale (1=no problem to 5=extreme problems). Change from baseline is being presented for EQ Index score. Index score is defined as a weighted combination of the levels of the 5-dimention scales, ranging from 0 to 1 (perfect health), with higher scores indicating better health-related quality of life. The United States value set from Pickard et al 2019 was used.
Time Frame: Baseline, every 3 cycles up to C48D1 (1 cycle = 28 days)
Population: FAS population with non-missing baseline EQ-5D-5L assessments. For each post-baseline timepoint, FAS population with non-missing baseline and post-baseline EQ-5D-5L assessment. FAS comprised of all patients to whom study treatment had been assigned by randomization.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 238 | 245
Scores on a scale
  Baseline (BL) | 0.78 (0.204) | 0.78 (0.239)
  Change from BL at Cycle (C) 3 Day (D) 1: number analyzed (Participants) | 205 | 199
  Change from BL at Cycle (C) 3 Day (D) 1 | 0.00 (0.215) | -0.03 (0.222)
  Change from BL at C6D1: number analyzed (Participants) | 163 | 157
  Change from BL at C6D1 | -0.02 (0.260) | -0.02 (0.305)
  Change from BL at C9D1: number analyzed (Participants) | 129 | 117
  Change from BL at C9D1 | 0.03 (0.232) | -0.01 (0.226)
  Change from BL at C12D1: number analyzed (Participants) | 93 | 88
  Change from BL at C12D1 | 0.02 (0.163) | -0.05 (0.261)
  Change from BL at C15D1: number analyzed (Participants) | 84 | 61
  Change from BL at C15D1 | -0.02 (0.238) | 0.01 (0.221)
  Change from BL at C18D1: number analyzed (Participants) | 65 | 53
  Change from BL at C18D1 | -0.02 (0.208) | 0.00 (0.226)
  Change from BL at C21D1: number analyzed (Participants) | 47 | 45
  Change from BL at C21D1 | 0.00 (0.208) | 0.00 (0.256)
  Change from BL at C24D1: number analyzed (Participants) | 45 | 41
  Change from BL at C24D1 | 0.00 (0.157) | 0.02 (0.225)
  Change from BL at C27D1: number analyzed (Participants) | 34 | 35
  Change from BL at C27D1 | -0.09 (0.283) | 0.00 (0.213)
  Change from BL at C30D1: number analyzed (Participants) | 30 | 25
  Change from BL at C30D1 | -0.03 (0.315) | 0.02 (0.256)
  Change from BL at C33D1: number analyzed (Participants) | 22 | 22
  Change from BL at C33D1 | -0.01 (0.211) | -0.02 (0.218)
  Change from BL at C36D1: number analyzed (Participants) | 18 | 15
  Change from BL at C36D1 | -0.07 (0.333) | -0.07 (0.395)
  Change from BL at C39D1: number analyzed (Participants) | 14 | 10
  Change from BL at C39D1 | -0.16 (0.360) | 0.02 (0.143)
  Change from BL at C42D1: number analyzed (Participants) | 9 | 4
  Change from BL at C42D1 | -0.09 (0.262) | -0.13 (0.309)
  Change from BL at C45D1: number analyzed (Participants) | 6 | 2
  Change from BL at C45D1 | -0.12 (0.262) | 0.17 (0.069)
  Change from BL at C48D1: number analyzed (Participants) | 1 | 2
  Change from BL at C48D1 | -0.07 (0.000) | 0.06 (0.087)

18. Secondary Outcome: Change From Baseline in the European Quality of Life (EuroQoL) - 5 Dimensions, 5 Level Questionnaire (EQ-5D-5L) Visual Analogue Scale (VAS) Over Time
Description: The EQ-5D-5L VAS records the participant's self-rated health on a visual analogue scale numbered from 0 to 100, with 0 being "the worst health you can imagine" and 100 being "the best health you can imagine". Change from baseline was presented.
Time Frame: Baseline, every 3 cycles up to C48D1 (1 cycle = 28 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 238 | 245
Scores on a scale
  Baseline (BL) | 68.91 (18.371) | 68.04 (18.762)
  Change from BL at Cycle 3 Day 1 (C3D1): number analyzed (Participants) | 205 | 199
  Change from BL at Cycle 3 Day 1 (C3D1) | 1.39 (21.029) | 0.40 (18.767)
  Change from BL at C6D1: number analyzed (Participants) | 163 | 157
  Change from BL at C6D1 | 2.60 (25.218) | 2.08 (23.294)
  Change from BL at C9D1: number analyzed (Participants) | 129 | 117
  Change from BL at C9D1 | 5.28 (20.528) | 2.55 (20.805)
  Change from BL at C12D1: number analyzed (Participants) | 93 | 88
  Change from BL at C12D1 | 5.55 (21.380) | 1.18 (22.728)
  Change from BL at C15D1: number analyzed (Participants) | 84 | 61
  Change from BL at C15D1 | 2.87 (21.940) | 3.72 (21.564)
  Change from BL at C18D1: number analyzed (Participants) | 65 | 53
  Change from BL at C18D1 | 3.80 (20.474) | 6.87 (19.369)
  Change from BL at C21D1: number analyzed (Participants) | 47 | 45
  Change from BL at C21D1 | 3.70 (23.541) | 5.71 (18.577)
  Change from BL at C24D1: number analyzed (Participants) | 45 | 41
  Change from BL at C24D1 | 1.73 (21.288) | 7.68 (18.781)
  Change from BL at C27D1: number analyzed (Participants) | 34 | 35
  Change from BL at C27D1 | -0.44 (21.139) | 4.63 (19.792)
  Change from BL at C30D1: number analyzed (Participants) | 30 | 25
  Change from BL at C30D1 | 3.13 (26.829) | 4.76 (14.998)
  Change from BL at C33D1: number analyzed (Participants) | 22 | 22
  Change from BL at C33D1 | 5.41 (26.923) | 1.64 (17.705)
  Change from BL at C36D1: number analyzed (Participants) | 18 | 15
  Change from BL at C36D1 | -1.50 (25.714) | -2.80 (29.617)
  Change from BL at C39D1: number analyzed (Participants) | 14 | 10
  Change from BL at C39D1 | 3.57 (28.281) | 1.70 (20.078)
  Change from BL at C42D1: number analyzed (Participants) | 9 | 4
  Change from BL at C42D1 | -11.89 (22.469) | -0.75 (26.550)
  Change from BL at C45D1: number analyzed (Participants) | 6 | 2
  Change from BL at C45D1 | 2.00 (15.113) | -2.00 (24.042)
  Change from BL at C48D1: number analyzed (Participants) | 1 | 2
  Change from BL at C48D1 | 7.00 (0.000) | 5.50 (34.648)

19. Secondary Outcome: Change From Baseline of Global Health Status/Quality of Life Scores Using European Organization for Research and Treatment of Cancer's Core Quality of Life Questionnaire (EORTC-QLQ-C30).
Description: EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer participants. Participant's responses to 2 questions (Items 29+30: "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall outcome. Change from baseline to Cycle 12 Day 1 as presented.
Time Frame: Up to Cycle 12 Day 1 (C12D1) (1 cycle = 28 days)
Population: FAS population with non-missing baseline (Cycle 1 Day 1) and Cycle 12 Day 1 EORTC-QLQ-C30 assessments. FAS comprised of all patients to whom study treatment had been assigned by randomization.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 64 | 62
Scores on a scale | 8.72 (23.071) | 8.20 (19.932)

20. Post Hoc Outcome: All Collected Deaths
Description: Deaths were collected from randomization until the end of the trial, approx. 52 months, including post-treatment survival follow up period.
Time Frame: from randomization until end of trial, up to approx. 52 months
Population: Clinical database population: All randomized participants: participants who died before treatment, during treatment and post-treatment.
Measure: Number; unit: Participants
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 265 | 265
Participants
  Pre-treatment deaths | 0 | 1
  On-treatment deaths | 18 | 37
  Post-treatment deaths: number analyzed (Participants) | 247 | 228
  Post-treatment deaths | 143 | 122
  All deaths | 161 | 160

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from the date of first administration of study treatment to 30 days after the date of the last administration of study treatment, up to maximum duration of 43.5 months (sabatolimab plus AZA) and 42.6 months (placebo + AZA). Deaths were collected from randomization until end of trial, approx. 52 months.
Description: Adverse Event: Any sign or symptom that occurs during the study treatment + 30 days post treatment. All-Cause Mortality is based on all randomized participants (by randomized study treatment), Serious and Other Adverse Events are summarized for the participants who received study treatment (by study treatment received).
Arm/Group | Sabatolimab (MBG453) + Azacitidine | Placebo + Azacitidine
All-Cause Mortality (participants affected / at risk) | 161/265 | 160/265
Serious Adverse Events (participants affected / at risk) | 174/263 | 164/265
Other Adverse Events (participants affected / at risk) | 256/263 | 255/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sabatolimab (MBG453) + Azacitidine (N=263) | Placebo + Azacitidine (N=265)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 3
Anaemia (Blood and lymphatic system disorders) | 11 | 11
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 1
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 49 | 31
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Myelosuppression (Blood and lymphatic system disorders) | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 4 | 1
Pancytopenia (Blood and lymphatic system disorders) | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 2
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 1
Atrial flutter (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 6 | 2
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Haematotympanum (Ear and labyrinth disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric dysplasia (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 3
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Melaena (Gastrointestinal disorders) | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0
Overflow diarrhoea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders and administration site conditions) | 1 | 1
Chest discomfort (General disorders and administration site conditions) | 1 | 0
Chest pain (General disorders and administration site conditions) | 2 | 0
Fatigue (General disorders and administration site conditions) | 1 | 0
General physical health deterioration (General disorders and administration site conditions) | 2 | 2
Multiple organ dysfunction syndrome (General disorders and administration site conditions) | 1 | 1
Oedema (General disorders and administration site conditions) | 1 | 0
Pain (General disorders and administration site conditions) | 1 | 0
Peripheral swelling (General disorders and administration site conditions) | 1 | 0
Pyrexia (General disorders and administration site conditions) | 17 | 19
Sudden death (General disorders and administration site conditions) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 6 | 1
Appendicitis (Infections and infestations) | 2 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 3
Bacterial infection (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 12 | 9
COVID-19 pneumonia (Infections and infestations) | 4 | 9
Candida infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 6 | 1
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 4 | 1
Encephalitis viral (Infections and infestations) | 0 | 1
Enterococcal sepsis (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 1
Eyelid infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 2
Herpes dermatitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 3
Legionella infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 5 | 2
Opportunistic infection (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 0 | 1
Periodontitis (Infections and infestations) | 0 | 1
Periorbital cellulitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 35 | 36
Pneumonia aspiration (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia escherichia (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Pulmonary mucormycosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 1 | 0
Renal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 3
Rhinovirus infection (Infections and infestations) | 2 | 0
Rotavirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 10
Septic shock (Infections and infestations) | 6 | 8
Sialoadenitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 2 | 2
Soft tissue infection (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 2
Systemic infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Urinary tract infection (Infections and infestations) | 7 | 5
Urinary tract infection enterococcal (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 1 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Refractoriness to platelet transfusion (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Stoma site inflammation (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 4 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Anti-platelet antibody positive (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 4 | 1
Ejection fraction decreased (Investigations) | 1 | 0
Liver function test increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 5 | 2
Platelet count decreased (Investigations) | 10 | 7
Transaminases increased (Investigations) | 1 | 0
Troponin T increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 1
Central nervous system haemorrhage (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Orthostatic intolerance (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 1 | 2
Confusional state (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 5
Calculus bladder (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal cyst haemorrhage (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Arterial thrombosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
White coat hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sabatolimab (MBG453) + Azacitidine (N=263) | Placebo + Azacitidine (N=265)
Anaemia (Blood and lymphatic system disorders) | 107 | 91
Febrile neutropenia (Blood and lymphatic system disorders) | 19 | 21
Leukopenia (Blood and lymphatic system disorders) | 17 | 22
Neutropenia (Blood and lymphatic system disorders) | 96 | 76
Thrombocytopenia (Blood and lymphatic system disorders) | 67 | 58
Abdominal pain (Gastrointestinal disorders) | 26 | 15
Constipation (Gastrointestinal disorders) | 141 | 114
Diarrhoea (Gastrointestinal disorders) | 61 | 46
Nausea (Gastrointestinal disorders) | 87 | 66
Stomatitis (Gastrointestinal disorders) | 14 | 12
Vomiting (Gastrointestinal disorders) | 48 | 45
Asthenia (General disorders and administration site conditions) | 31 | 29
Fatigue (General disorders and administration site conditions) | 50 | 33
Injection site reaction (General disorders and administration site conditions) | 16 | 20
Oedema peripheral (General disorders and administration site conditions) | 24 | 33
Pyrexia (General disorders and administration site conditions) | 71 | 59
COVID-19 (Infections and infestations) | 44 | 35
Cellulitis (Infections and infestations) | 14 | 12
Pneumonia (Infections and infestations) | 30 | 27
Upper respiratory tract infection (Infections and infestations) | 21 | 20
Urinary tract infection (Infections and infestations) | 24 | 17
Fall (Injury, poisoning and procedural complications) | 15 | 5
Alanine aminotransferase increased (Investigations) | 15 | 24
Aspartate aminotransferase increased (Investigations) | 12 | 18
Blood creatinine increased (Investigations) | 19 | 12
C-reactive protein increased (Investigations) | 18 | 6
Lymphocyte count decreased (Investigations) | 14 | 20
Neutrophil count decreased (Investigations) | 61 | 54
Platelet count decreased (Investigations) | 62 | 56
Weight decreased (Investigations) | 34 | 25
White blood cell count decreased (Investigations) | 48 | 52
Decreased appetite (Metabolism and nutrition disorders) | 26 | 26
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 25
Hyperuricaemia (Metabolism and nutrition disorders) | 16 | 18
Hypoalbuminaemia (Metabolism and nutrition disorders) | 20 | 23
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 15
Hypokalaemia (Metabolism and nutrition disorders) | 39 | 33
Hyponatraemia (Metabolism and nutrition disorders) | 15 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 43 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 9
Dizziness (Nervous system disorders) | 21 | 15
Headache (Nervous system disorders) | 23 | 20
Insomnia (Psychiatric disorders) | 29 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 18
Rash (Skin and subcutaneous tissue disorders) | 30 | 26
Hypertension (Vascular disorders) | 21 | 12
Hypotension (Vascular disorders) | 17 | 14

LIMITATIONS AND CAVEATS:
A total of 530 participants were randomized (265 to sabatolimab+AZA, 265 to placebo+AZA), but 1 participant in each arm did not receive any study treatment and were excluded from the Safety Set. Another sabatolimab-assigned participant received only AZA and thus was summarized in the placebo+AZA arm in all safety analyses. Therefore, the Serious and Other Adverse Events were shown for 263 sabatolimab+AZA and 265 placebo+AZA participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of pooled data (i.e. data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT04266301/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT04266301/SAP_001.pdf